CLINICAL TRIAL: NCT04987580
Title: Efficacy and Safety of a Single Syringe Total Intravenous Anesthesia With Propofol and Remifentanil: A Prospective Cohort Study
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: Single Syringe TIVA
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this prospective observational study was to evaluate the efficacy and safety of single syringe TIVA with propofol and remifentanil. The primary outcome for efficacy was a processed EEG (pEEG) index within the recommended range for general anesthesia for the duration of the maintenance anesthetic. The primary outcome measure for safety was intraoperative administration of vasopressors. We hypothesized that the pEEG index would be within the recommended range for over 90% of the duration of the maintenance anesthetic. We hypothesized that vasopressor use would be consistent with other anesthetic types using potent inhaled agents.

DETAILED DESCRIPTION:
Total intravenous anesthesia (TIVA) is a commonly used general anesthetic. Propofol and remifentanil is a common drug combination used in TIVA and is a safe and efficacious method of anesthesia in pediatric and adult patients.[1-7] A typical TIVA method is to administer each drug using a separate syringe pump. Another approach to TIVA is to use a single syringe pump containing propofol and remifentanil. This approach is considered off-label as neither drug has been approved by a national or international regulatory agency to be used in a single syringe.

The efficacy and safety of single syringe TIVA has not yet been evaluated. At a single university hospital center, single syringe TIVA with propofol and remifentanil has been used for over 15 years for a variety of procedures. A common combination of propofol and remifentanil in a single syringe is propofol 10 mg/ml and remifentanil 20 mcg/ml.

A preliminary retrospective analysis of electronic medical records (Epic Hyperspace Electronic Medical Record, Epic Systems Corporation, Verona, Wisconsin) from May of 2014 to June of 2019 identified 21,985 procedures using single syringe TIVA. (unpublished data) This retrospective analysis, was used to identify adverse events, which included: awareness during surgery, significant vasopressor use, replacement of the single syringe TIVA with an inhaled anesthetic, and patient injury or death. This analysis was limited by possible clinician underreporting of vasopressor use, changes in TIVA infusion rates, and awareness events.

The purpose of this prospective observational study was to evaluate the efficacy and safety of single syringe TIVA with propofol and remifentanil. The primary outcome for efficacy was a processed EEG (pEEG) index within the recommended range for general anesthesia for the duration of the maintenance anesthetic. The primary outcome measure for safety was intraoperative administration of vasopressors. We hypothesized that the pEEG index would be within the recommended range for over 90% of the duration of the maintenance anesthetic. We hypothesized that vasopressor use would be consistent with other anesthetic types using potent inhaled agents.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 75
* Elective orthopedic surgery patients for whom the use of propofol (10 mg/ml) in combination with remifentanil (20 mcg/ml) used in a single syringe in indicated

Exclusion Criteria:

* True allergy to propofol/remifentanil
* Inability to understand pain scores and other questionnaires
* Inability to speak English
* Emergency surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to an orthopedic surgery center for elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of Single Syringe TIVA | during the surgery
  Duration of time that processed EEG values are within acceptable limits during maintenance of anesthesia

SECONDARY OUTCOMES:
Hemodynamic Instability | during the surgery
  Blood pressure readings will be recorded
Incidence of vasoactive dosage | during the surgery
  Vasoactive agent use will be recorded
Intra-operative movement | during the surgery
  Intra-operative movement will be recorded during the surgery
Time to emergence | during the surgery
  Time to emergence from anesthesia will be recorded during the surgery
Anesthesia provider team | Immediately following the surgery
  Anesthesia provider(s) (i.e. anesthetist attending, CRNA, resident) will be recorded.
Post-operative nausea | 0, 15, 30, and 45 minutes after the surgery
  Post-operative nausea will be recorded
Post-operative vomiting | 0, 15, 30, and 45 minutes after the surgery
  Post-operative vomiting will be recorded
Awareness with recall | 30 minutes and 1 day after the surgery
  Awareness will be assessed using the structured interview
Post-operative delirium | 45 minutes after the surgery
  Post-operative delirium will be recorded using the Nursing Delirium Screening Scale (0-mild (positive outcome), 1-moderate, 2-severe (poor outcome)).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States